CLINICAL TRIAL: NCT06943456
Title: Comparison of Outcome of Open Appendectomy With and Without Transversus Abdominis Plane Block
Brief Title: Comparison of Outcome of Open Appendectomy With and Without Transversus Abdominis Plane (TAP) Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Hafiz Rana Kamran Ijaz, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exp131
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Appendicitis; Postoperative Pain
MeSH Terms: conditions — Appendicitis; Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups:
  Group A will receive a Transversus Abdominis Plane (TAP) block following open appendectomy.
  Group B will undergo the same surgical procedure without a TAP block.
  Each group will receive only one type of intervention, and both will be observed independently for outcomes such as postoperative pain, complications, and hospital stay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Appendectomy with Transversus Abdominis Plane (TAP) Block (Experimental): Patients in this group will undergo open appendectomy followed by the administration of a Transversus Abdominis Plane (TAP) block. The TAP block will be performed using a mixture of 10 ml of 1% lignocaine and 10 ml of 0.5% bupivacaine, injected between the transversus abdominis and internal oblique muscles under vision. This intervention is designed to provide localized post-operative analgesia and reduce the need for systemic opioid analgesics.
  Interventions: Procedure: Transversus Abdominis Plane (TAP) Block for Postoperative Pain Management
- Open Appendectomy without Transversus Abdominis Plane (TAP) Block (Active Comparator): Patients in this group will undergo open appendectomy using the standard surgical technique without the administration of a Transversus Abdominis Plane (TAP) block. Post-operative pain will be managed using standard opioid analgesia as required, without the benefit of the TAP block for localized pain relief.
  Interventions: Procedure: Standard Open Appendectomy with Postoperative Pain Management

INTERVENTIONS:
Procedure: Transversus Abdominis Plane (TAP) Block for Postoperative Pain Management — The intervention involves the administration of a Transversus Abdominis Plane (TAP) block performed at the end of an open appendectomy surgery. A mixture of 10 ml of 1% lignocaine and 10 ml of 0.5% bupivacaine is injected into the transversus abdominis plane, located between the transversus abdominis and internal oblique muscles, under direct vision. This procedure aims to provide localized pain relief by blocking the sensory nerves of the anterior abdominal wall, reducing the need for systemic opioid analgesics during post-operative recovery
  Arms: Open Appendectomy with Transversus Abdominis Plane (TAP) Block
Procedure: Standard Open Appendectomy with Postoperative Pain Management — The intervention involves the standard open appendectomy surgical procedure without the addition of a Transversus Abdominis Plane (TAP) block. Postoperative pain management in this group is managed using standard opioid analgesics. No local anesthetic block is performed, and pain management is entirely reliant on systemic medications, including opioids, for post-operative recovery
  Arms: Open Appendectomy without Transversus Abdominis Plane (TAP) Block

SUMMARY:
This study is being conducted to compare two types of pain management techniques in patients undergoing open appendectomy (surgical removal of the appendix through a traditional incision).

One group of patients will receive a Transversus Abdominis Plane (TAP) block, a type of regional anesthesia given at the end of surgery to numb the abdominal area and reduce pain. The other group will undergo the same surgery without receiving the TAP block.

The purpose of this study is to find out whether adding the TAP block helps in:

Reducing postoperative pain

Shortening the hospital stay

Minimizing complications like nausea, vomiting, and delayed mobility

Improving patient satisfaction after surgery

Opioid medications are commonly used for pain control after surgery, but they come with side effects such as nausea, vomiting, dizziness, and risk of dependency. TAP block offers a promising alternative that may reduce or eliminate the need for opioids by targeting specific nerves in the abdominal wall.

This will be a randomized controlled trial (considered the gold standard in medical research), meaning patients will be randomly assigned to one of the two groups to ensure fair comparison. The study will enroll 136 adult patients who are diagnosed with appendicitis and are scheduled for open appendectomy at Jinnah Hospital Lahore.

By conducting this study, the researchers aim to provide strong scientific evidence on whether TAP block should be routinely used in appendectomy patients to enhance recovery and comfort. If proven effective, this could influence hospital protocols and improve post-surgery care both locally and internationally.

DETAILED DESCRIPTION:
Open appendectomy is one of the most frequently performed emergency surgeries worldwide for the treatment of acute appendicitis. Postoperative pain following this surgery can delay recovery, prolong hospital stay, and increase the risk of complications such as respiratory distress and venous thromboembolism due to reduced mobility.

Traditionally, postoperative pain is managed using systemic analgesics, particularly opioids. However, opioids are associated with significant side effects such as nausea, vomiting, respiratory depression, gastrointestinal disturbances, dizziness, urinary retention, and risk of dependence. This has prompted the search for safer and more effective alternatives, especially in resource-limited settings.

The Transversus Abdominis Plane (TAP) block is a regional anesthesia technique that involves the injection of local anesthetics into the fascial plane between the internal oblique and transversus abdominis muscles. This approach targets the sensory nerves supplying the anterior abdominal wall (T6-L1), providing effective somatic pain relief.

Several international studies have indicated that TAP block can significantly reduce postoperative pain scores and opioid consumption, particularly in abdominal surgeries. However, most of these studies are either retrospective or conducted outside the local context. In Pakistan, limited data exists, and the use of TAP block is not yet widespread or standardized in clinical practice.

This randomized controlled trial (RCT) is designed to evaluate the efficacy of TAP block in adult patients undergoing open appendectomy at Jinnah Hospital, Lahore. The study will enroll 136 participants, who will be randomized into two equal groups:

Group A will receive a TAP block with 10 ml of 1% lignocaine and 10 ml of 0.5% bupivacaine administered under direct vision at the end of the surgery.

Group B will undergo the same surgical procedure without the TAP block.

All surgeries will follow a standardized open appendectomy technique using a gridiron or Lanz incision. The TAP block will be performed in the midaxillary line between the anterior superior iliac spine and the subcostal margin under direct vision.

Pain will be assessed using the Visual Analog Scale (VAS) at multiple time points postoperatively (12, 16, and 24 hours). Additional parameters such as duration of hospital stay, postoperative complications (e.g., nausea, vomiting, delayed mobilization), and overall patient satisfaction will also be recorded.

The results from this study will help determine whether TAP block should be recommended as part of standard postoperative analgesia for open appendectomy. If the TAP block is found to be effective, it may reduce reliance on opioids, improve recovery times, and enhance patient outcomes-supporting broader implementation in surgical practices, especially in public-sector hospitals across developing regions.

This study adheres to ethical standards, with approval from the institutional ethical review committee, and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Both male and female patients.
* Patients fit for general anesthesia.
* Clinical findings of appendicitis.
* Lower right quadrant or periumbilical pain radiating to the right lower quadrant, with nausea and/or vomiting.
* Fever >38°C.
* Tenderness with Alvarado score >7.

Exclusion Criteria:

* Duration of symptoms >5 days.
* Absence of clinical findings of appendicitis.
* Palpable mass on physical examination suspected for appendiceal abscess.
* History of cirrhosis or hematological disorders.
* Allergic to or contraindicated for general anesthesia.
* Pregnancy.
* Patients who do not consent to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 12, 16, and 24 hours post-surgery
  Postoperative pain will be measured using the Visual Analog Scale (VAS) at 12, 16, and 24 hours post-surgery. The VAS is a scale where 0 represents no pain and 10 represents the worst possible pain. Patients will mark their pain intensity on a 10 cm line, and the score is measured by the distance (in centimeters) from the 'no pain' mark to the point marked by the patient. This scale provides a continuous variable to assess pain intensity, allowing a detailed understanding of pain levels over time. The VAS score will be used to compare the pain outcomes between the two groups (TAP block versus no TAP block).

IPD SHARING:
Plan to Share IPD: Undecided